CLINICAL TRIAL: NCT03564652
Title: Nutritional Support for Lactating Women and Azithromycin to Infants to Improve Growth Outcomes in Peri-urban Slums of Karachi, Pakistan - Randomized Controlled Trial
Brief Title: Nutritional Support for Lactating Women and Azithromycin to Infants - Mumta Lactating Women Trial
Acronym: MumtaLW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vital Pakistan Trust (Other)
Collaborators: Aga Khan University (Other)
Responsible Party: Principal Investigator, Yasir Shafiq, Research Manager, Vital Pakistan Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 002-VPT-IRB-18
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Undernutrition
MeSH Terms: conditions — Malnutrition | interventions — Azithromycin; Suspensions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (No Intervention): Control arm: Lactating women (LW) randomized in this arm will only receive standard of care which comprises of standard nutritional counseling, key messages of exclusive breastfeeding, essential newborn and infant care and immunization.
- Arm B (Experimental): Intervention arm B: Lactating women (LW) randomized in this arm will receive ready-to-use nutritional supplement, 'Balanced energy-protein (BEP)' for next 6 months to be consumed in a dose of 2 sachets of 75 grams per day. Further, LW will also receive standard of care which comprises of standard nutritional counseling, key messages of exclusive breastfeeding, essential newborn and infant care and immunization.
  Interventions: Dietary Supplement: Balanced energy-protein (BEP)
- Arm C (Experimental): Intervention arm B: Lactating women (LW) randomized in this arm will receive ready-to-use nutritional supplement, 'Balanced energy-protein (BEP)' for next 6 months to be consumed in a dose of 2 sachets of 75 grams per day. Further, the same infant of LW will receive a single dose of Azithromycin (20mg/kilogram) at day 42 of age. Further, LW will also receive standard of care which comprises of standard nutritional counseling, key messages of exclusive breastfeeding, essential newborn and infant care and immunization.
  Interventions: Dietary Supplement: Balanced energy-protein (BEP); Drug: Azithromycin

INTERVENTIONS:
Dietary Supplement: Balanced energy-protein (BEP) — Lactating women in the intervention arms will receive approximately 800 Kcal/day and around 16-21 gram of protein in a day in the form of ready-to-use supplement.
  Other Names: RUSF
  Arms: Arm B; Arm C
Drug: Azithromycin — A single prophylaxis dose of 20 mg/kg in suspension form, reconstituted by trial staff before dose administration by the same.
  Other Names: Suspension
  Arms: Arm C

SUMMARY:
A community-based, randomized control, assessor blinded trial in peri-urban settings of Karachi, Pakistan to study the impact of Lipid-based Nutritional Supplement for Pregnant and Lactating women which is balanced energy-protein (BEP) dietary supplement, a locally produced ready-to-use nutritional product for lactating women (LW) and single prophylaxis dose of Azithromycin for infants, on growth of infants over the period of six months since birth compared to current standard of care. LW and her infant will be enrolled in the trial within 168 hours of the birth and LW will be randomized in either of the arm:

1. Arm A: 'Control Arm', LW will only receive standard of care which comprises of standard nutritional counseling, key messages of exclusive breastfeeding, essential newborn and infant care and immunization.
2. Arm B: 'Nutritional supplement only', LW randomized will recieve nutrition supplement product for next 6 months to be consumed in a dose of 2 sachets of 75 grams per day. Further, LW will also receive standard of care which comprises of standard nutritional counseling, key messages of exclusive breastfeeding, essential newborn and infant care and immunization.
3. Arm C: ''Nutritional supplement plus Azithromycin', LW randomized will receive nutritional supplement product for next 6 months to be consumed in a dose of 2 sachets of 75 grams per day. Further, the infant of LW will receive a single dose of Azithromycin (20mg/kilogram) at day 42 of age. Further, LW will also receive standard of care which comprises of standard nutritional counseling, key messages of exclusive breastfeeding, essential newborn and infant care and immunization.

Study aim is to assess the efficacy of nutritional product in a proposed dose to lactating women for at least 6 months of lactation, alone or in combination of single dose of Azithromycin as 20mg/kg to infants at 42 days of age on lenght velocity as primary, and weight velocity as secondary outcome.

Participants will receive nutrition counseling along with guidance related to exclusive breastfeeding and further assessment will be done to assess breast milk composition, Haemoglobin, Ferritin and Transferrin receptor, and inflammatory biomarkers, as secondary outcomes. Further, this study will also look at the comparison of length-for-age, weight-for-length, and weight-for-age Z scores as other secondary outcome at 6 months of age among three arms.

ELIGIBILITY:
Inclusion Criteria:

* Mid-upper-arm-circumference of lactating women less than 23.0 cm, whose birth outcome should be captured within 168 hours
* Singleton alive baby
* Intention to stay in the catchment area for the entire duration of the trial after enrolment
* Intention to breastfeed the child for at least 6 months
* Voluntary written consent

Exclusion Criteria:

* Weight of newborn at first assessment, within 168 hours of birth is less than 1500 gm
* Newborn with known congenital anomaly or sign of serious illness based of study physician's assessment before enrollment.
* Lactating women has known allergies to peanut, lentils, chickpea or dairy products.
* Lactating woman who have some serious medical illness/condition due to which she is not able to or not willing to breastfeed the child, like breast cancer, inverted nipples.
* Previous enrolment in the same trial.

Ages: 13 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Lactating women
Enrollment: 957 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Length velocity at 6 months of infant's age | 6 months of infant age, after birth and enrollment through monthly assessment
  Mean difference in length velocity of >0.12 cm /month to look at comparisons between multiple arms

SECONDARY OUTCOMES:
Growth velocity at 6 months of infant's age | 6 months of infant age, after birth and enrollment through monthly assessment
  Mean difference in growth velocity of >0.4 gram/kg/day to look at comparisons between multiple arms
Length-for-Age Z-score (LAZ) of infants at 6 months of age | 6 months of infant age, after birth and enrollment through monthly assessment
  Mean difference in LAZ >0.5 to look at comparisons between multiple arms
Weight-for-Length Z-score (WLZ) of infants at 6 months of age | 6 months of infant age, after birth and enrollment through monthly assessment
  Mean difference in WLZ of >0.5 to look at comparisons between multiple arms
Weight-for-Age Z-score of (WAZ) infants at 6 months of age | 6 months of infant age, after birth and enrollment through monthly assessment
  Mean difference in WAZ of >0.5 to look at comparisons between multiple arms

OTHER OUTCOMES:
Breast milk composition | breast milk specimens will be collected at day 40-42 and 56 of infant age
  50 systematically selected lactating women in each arm will be approached for breast milk specimen to assess quality of breast milk composition (macro- and micro-nutrients), Human Milk Oligosaccharides (HMO), immunoglobulins and microbiome analysis. Same 50 women will be selected for outcome 7 and 8
Stool specimens of lactating women and infants | At day 40-42 and 56 of infant age
  Same 50 systematically selected lactating women in each arm will also be approached for stool samples on the same day and stool from the same infant will also be collected. Stool will be collected for TaqMan Array Card (TAC) analysis of enteric pathogens, B. Infantis, Calprotectin, Lipocalin 2 and Myeloperoxidase (MPO) as a marker of gut inflammation and will be assessed using a metagenomic approach
Blood specimens of lactating women | At day 40-42 and 56 of infant age
  Same 50 systematically selected lactating women in each arm will be approached for blood specimens to assess haemoglobin, serum Ferritin, Transferrin receptor and Acute phase proteins such as AGP and CRP
Blood specimens of infants | At day 40-42 and 56 of infant age
  All infants will be approached for blood speciemens to assess haemoglobin, serum Ferritin, Transferrin receptor, plasma proteomics and Acute phase proteins such as AGP and CRP

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Shafiq, MSc, Principal Investigator — Vital Pakistan Trust
Locations (1):
- Peri-urban slums of Karachi (Rehri Goth, Bhains Colony and Ali Akber Shah Goth), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Muhammad A, Shafiq Y, Nisar MI, Baloch B, Pasha A, Yazdani NS, Rizvi A, Muhammad S, Jehan F. Effect of maternal postnatal balanced energy protein supplementation and infant azithromycin on infant growth outcomes: an open-label randomized controlled trial. Am J Clin Nutr. 2024 Sep;120(3):550-559. doi: 10.1016/j.ajcnut.2024.06.008. Epub 2024 Jun 24. PMID 38925354
- [Derived] Muhammad A, Shafiq Y, Nisar MI, Baloch B, Yazdani AT, Yazdani N, Jehan F. Nutritional support for lactating women with or without azithromycin for infants compared to breastfeeding counseling alone in improving the 6-month growth outcomes among infants of peri-urban slums in Karachi, Pakistan-the protocol for a multiarm assessor-blinded randomized controlled trial (Mumta LW trial). Trials. 2020 Sep 1;21(1):756. doi: 10.1186/s13063-020-04662-y. PMID 32873314

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-11-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT03564652/SAP_000.pdf
  • Study Protocol (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT03564652/Prot_001.pdf